CLINICAL TRIAL: NCT00834808
Title: A Dose Linearity Study of the Labopharm Formulation of Tramadol HCl/Contramid®, 100 mg, 200 mg and 300 mg After A Single Oral Administration In Fasting Condition, In Healthy Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Vice-President Regulatory Affairs, Labopharm Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MDT1-011
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Tramadol

ARMS (3):
- 1: Tramadol HCl 100mg (Experimental)
  Interventions: Drug: Tramadol HCl
- 2: Tramadol HCl 200mg (Experimental)
  Interventions: Drug: Tramadol HCl
- 3: Tramadol HCl 300mg (Experimental)
  Interventions: Drug: Tramadol HCl

INTERVENTIONS:
Drug: Tramadol HCl — One single oral administration of Tramadol HCl 100 mg, 200 mg or 300 mg as per randomization schedule.

SUMMARY:
The purposes of this study were:

* To evaluate the plasma pharmacokinetic profile of tramadol and its principal metabolite, the O-desmethyltramadol, after a single oral administration of 100, 200 and 300 mg of tramadol as the Labopharm extended-release formulation prepared with Contramid.
* To assess the dose linearity of tramadol and its principal metabolite, the O-desmethyltramadol, between 100 mg and 300 mg following a single dose administration of the Labopharm extended-release formulation prepared with Contramid under fasting conditions in young healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form duly signed by the subject.
* Males aged from 18 to 45 years inclusively and with Body Mass Index (BMI) between 18 and 30 kg/m2 inclusively.
* Clinical laboratory values within 10% above or below the laboratory's stated normal range; if not within this range, the clinical investigator will decide if they were not clinically significant and recorded this fact on the Case Report Form (CRF).
* Healthy according to the physical examination and laboratory results.
* Normal cardiovascular function according to a 12-lead electrocardiogram (ECG).
* Non-smoker or subjects smoking no more than 5 cigarettes per day (or equivalent) and able to abstain from smoking during inpatient phases of the study.
* Subjects covered by Social Security in compliance with the recommendations of French Law relating to biomedical research.
* Subjects with normal dietary requirements (neither vegetarian, nor on a diet).

Exclusion Criteria:

* History of hypersensitivity to tramadol or any other compounds.
* Presence or significant history of gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Presence or significant history of cardiovascular, pulmonary, haematological, neoplasic, neurological, psychiatric, endocrine, immunological or dermatological disease.
* Presence or significant history of glaucoma.
* Supine pulse rate lower than 45 beats per minute (bpm) after 5 minutes at rest or higher than 100 bpm.
* History of hypotensive episodes or a standing systolic blood pressure reading of <100 mmHg or a diastolic reading of <45 mmHg, measured on the screening day.
* History of hypertensive episodes or a supine systolic blood pressure reading of >145 mmHg or a diastolic reading of >95 mmHg, measured on the screening day.
* Presence of atrioventricular (AV) block assessed during pre-study evaluation or during the study. The lower limit considered for a first degree AV block was be a PR interval of 200 millisecond (msec).
* Maintenance therapy with any drug, or history of drug dependency, alcohol abuse (>3 units of alcohol per day), or serious psychological disease.
* Subjects consuming large quantities of drinks containing xanthine bases (coffee, tea, chocolate or cola; more than 6 cups or glasses per day).
* Any clinically significant illness in the previous 21 days before day 1 of this study.
* Subjects who had undergone general anesthesia within 3 months prior to the present study.
* Use of drugs known to affect liver enzymes (eg, inducers or inhibitors of Cytochrome P450) in the previous 30 days before day 1 of this study (eg, all barbiturates, corticosteroids, di & methyl-phenylhydantoin).
* Use of any medication (including OTC preparations) in the previous 14 days before day 1 of this study.
* Donation of 350 mL (or more) of blood in the previous 3 months or participation in another clinical trial in the previous 3 months before day 1 of this study.
* Subjects undergoing dental care.
* Positive urine drug screening.
* Positive results to human immunodeficiency virus (HIV) 1 & 2 or hepatitis B surface antigen (HBsAg) or anti-HCV (hepatitis C virus) tests.
* History of fainting upon blood sampling.
* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of the consent to participate in the study or to limit the ability to comply with the protocol requirements.
* Subjects unable to abstain from intensive muscular effort or sport competitions during the week prior to the study and throughout the study itself.
* Subjects who had forfeited his freedom by administrative or legal award or who were under guardianship.
* Subjects who received the ceiling amount of 25,000 francs within the last 12 months or who reached this ceiling with the payment of this allowance for this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2002-11; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

REFERENCES:
- [Result] Karhu D, El-Jammal A, Dupain T, Gaulin D, Bouchard S. Pharmacokinetics and dose proportionality of three Tramadol Contramid OAD tablet strengths. Biopharm Drug Dispos. 2007 Sep;28(6):323-30. doi: 10.1002/bdd.561. PMID 17575561
- See also: Approved labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=9048

RESULTS

PARTICIPANT FLOW:
Groups:
- 1: Tramadol HCl 100mg; 2: Tramadol HCl 200mg; 3: Tramadol HCl 300mg: * Single oral administration fasting conditions.
  * Randomization schedule based on a Latin Square design.
Period: Treatment Period 1 (Day 1)
Arm/Group | 1: Tramadol HCl 100mg | 2: Tramadol HCl 200mg | 3: Tramadol HCl 300mg
Started | 9 | 9 | 9
Completed | 9 | 9 | 9
Not Completed | 0 | 0 | 0
Period: Treatment Period 2 (Day 8)
Arm/Group | 1: Tramadol HCl 100mg | 2: Tramadol HCl 200mg | 3: Tramadol HCl 300mg
Started | 9 | 9 | 9
Completed | 9 | 9 | 9
Not Completed | 0 | 0 | 0
Period: Treatment Period 3 (Day 15)
Arm/Group | 1: Tramadol HCl 100mg | 2: Tramadol HCl 200mg | 3: Tramadol HCl 300mg
Started | 9 | 9 | 9
Completed | 9 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Tramadol HCl 100mg | 2: Tramadol HCl 200mg | 3: Tramadol HCl 300mg | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0.0
  Between 18 and 65 years | 9 | 9 | 9 | 27.0
  >=65 years | 0 | 0 | 0 | 0.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0.0
  Male | 9 | 9 | 9 | 27.0

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-t)
Description: Area under the plasma concentration versus time curve to the last measurable concentration.
  h = hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | 1: Tramadol HCl 100mg | 2: Tramadol HCl 200mg | 3: Tramadol HCl 300mg
Number analyzed (Participants) | 9 | 9 | 9
ng.h/mL | 2064 (707) | 4332 (1149) | 6568 (2050)

2. Primary Outcome: AUC(0-inf)
Description: Area under the plasma concentration versus time curve extrapolated to infinity. h = hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | 1: Tramadol HCl 100mg | 2: Tramadol HCl 200mg | 3: Tramadol HCl 300mg
Number analyzed (Participants) | 9 | 9 | 9
ng.h/mL | 2108 (731) | 4416 (1192) | 6741 (2156)

3. Primary Outcome: Cmax
Description: Maximum plasma concentration.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 1: Tramadol HCl 100mg | 2: Tramadol HCl 200mg | 3: Tramadol HCl 300mg
Number analyzed (Participants) | 9 | 9 | 9
ng/mL | 91 (27) | 197 (58) | 290 (147)

4. Secondary Outcome: Tmax
Description: Time to maximum plasma concentration
Time Frame: 48 hours
Measure: Median (Full Range); unit: hours
Arm/Group | 1: Tramadol HCl 100mg | 2: Tramadol HCl 200mg | 3: Tramadol HCl 300mg
Number analyzed (Participants) | 9 | 9 | 9
hours | 9 [3 to 16] | 5.5 [3 to 16] | 5 [3 to 24]

5. Secondary Outcome: t1/2
Description: Apparent terminal elimination half-life
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1: Tramadol HCl 100mg | 2: Tramadol HCl 200mg | 3: Tramadol HCl 300mg
Number analyzed (Participants) | 9 | 9 | 9
hours | 6.1 (1.3) | 6.1 (1.3) | 6.3 (1.5)

ADVERSE EVENTS:
Arm/Group | 1: Tramadol HCl 100mg | 2: Tramadol HCl 200mg | 3: Tramadol HCl 300mg
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publication of the results obtained will be authorized, after prior agreement between the various recipients [investigator and sponsor].